CLINICAL TRIAL: NCT00395291
Title: Growth Hormone Secretagogue MK-0677 Effect on IGF-1 Levels in ESRD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Warren K Bolton, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 12569
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-01

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease
Keywords: Chronic kidney disease; End stage renal disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — ibutamoren mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MK-0677 then Placebo (Experimental): MK-0677 and Placebo - All subjects were given MK-0677 for a 30 +/- 7 days and then they were given a placebo for 30 +/- 7 days.
  Interventions: Drug: MK-0677; Drug: Placebo
- Placebo then MK-0677 (Experimental): MK-0677 and Placebo - All subjects were given Placebo for a 30 +/- 7 days and then they were given MK-0677 for 30 +/- 7 days.
  Interventions: Drug: MK-0677; Drug: Placebo

INTERVENTIONS:
Drug: MK-0677 — The dosage of the drug is 25mg, subjects will take one pill a day for about 30 days.
Drug: Placebo — Placebo

SUMMARY:
The objective of this study is to determine MK-0677 increases IGF-1 in patients with end stage renal disease (ESRD) on hemodialysis.

DETAILED DESCRIPTION:
With development and progression of chronic kidney disease (CKD) to end stage renal disease (ESRD), malnutrition becomes an increasingly severe problem. This is thought to occur from two mechanisms: decreased appetite secondary to uremia and development of a catabolic inflammatory milieu. Patients experience decreased muscle mass and functional activity associated with increased morbidity and mortality. Many therapies to improve poor nutritional state have been used with little success. Growth hormone (GH) and insulin like growth hormone (IGF-1) improve muscle mass, quality of life, nutritional parameters, immune and physical functions but must be given parenterally and are limited by expense and patient compliance. Recently, the endogenous GH receptor secretagogue (GHRS) ghrelin has been shown to raise endogenous GH and improve food intake but must be given parenterally and is not available. The experimental drug MK-0677, a synthetic GHRS, ghrelin mimetic, which is given orally, has recently been shown to increase IGF-1 and muscle mass in the elderly. Its effects in CKD and ESRD are unknown. We will study the effects of MK-0677 on renal patients. Specifically, we hope to show that the drug increases IGF-1 in renal patients, and has similar effects to exogenous GH and IGF-1. Subjects will be ESRD hemodialysis patients. This protocol is an investigator-initiated, randomized, double-blind crossover, placebo-controlled pilot study. The study's primary outcome is IGF-1 levels for subjects. Secondary outcomes will be levels of cytokines, esterase, leptin, insulin, ghrelin, TNF-alpha, CRPs, IL-1, IL-6, IL-10, and adiponectin.

ELIGIBILITY:
Inclusion Criteria:

- GFR by the MDRD estimate < 30ml/minute/1.73m2 or on hemodialysis

Exclusion Criteria:

* Body mass index greater than 35 kg/m2, or morbid obesity
* Uncontrolled hypothyroidism, defined as an elevated serum thyroid stimulating hormone (THS) and a free serum thyroxine (T4) less than the lower limit of normal, when tested at baseline (Patients requiring thyroid replacement during the study may continue.)
* Uncontrolled hyperthyroidism, defined as a TSH less than the lower limit of normal and an elevated free T4, when tested at baseline
* Hemoglobin <10 Gm/dl
* Elevated serum transaminases (>2.0 times the upper limit of normal at baseline)
* Diabetes with one of more of the following:

  1. Poorly controlled diabetes as defined by a HbA1C > 7.0% at baseline)
  2. Proliferative diabetic retinopathy [To participate in this study, diabetic patients will need to have had a dilated ophthalmology exam within 12 months of enrollment. Individuals who already have extensive background retinopathy will need to have a dilated ophthalmology exam within the 3 months of enrollment. Patients with pre-proliferative or proliferative retinopathy will be excluded].
  3. Unwilling or unable to check blood glucose at home at least daily.
* Currently receiving a systemic corticosteroid dose of >10 mg prednisone (or equivalent), or patient has received, for a duration > 30 days in the previous 6 months (i.e., prior to signing the informed consent form), a systemic corticosteroid dose of > 10 mg prednisone (or equivalent). (The previous use, or current use, of a topical or inhaled corticosteroid is allowed.)
* Currently taking or previously on an anabolic steroid or growth hormone at any dose, or for any duration, during the 12 months prior to study entry.
* Significant end-organ disease, other than kidney disease, which, in the opinion of the investigator may pose an added risk to the patient, confound the study results, or impair the patient's ability to complete the trial.
* Any of the following disorders within 6 months prior to baseline:

  1. Acute coronary syndrome (e.g., myocardial infarction or unstable angina)
  2. Coronary artery intervention (e.g., coronary bypass graft [CABG], percutaneous transluminal coronary angioplasty [PTCA]).
  3. Stroke or transient ischemic neurological disorder (e.g. transient ischemic attack [TIA])
* New or worsening signs or symptoms of coronary heart disease within the 3 months prior to baseline.
* NYHA (New York Heart Association)Class III or IV congestive heart failure (definitions shown in Appendix A)
* Uncontrolled hypertension when checked at screening visit: as evidenced by > 160 systolic and/or 100 diastolic (measured in dominant or non-dialysis access arm, after at least 5 minutes, sitting)
* Cancer, or diagnosis of malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or adequately treated in situ cervical cancer.
* Active carpal tunnel syndrome
* Patient is, in the opinion of the investigator, mentally or legally incapacitated such that informed consent cannot be obtained or such that adherence to the study procedures and dosing regimens is questionable.
* Patient is, at study entry, a regular user (including "recreational use") of illicit drugs or had a recent history (within the last 5 years) of drug or alcohol abuse.
* Patient plans to relocate or change to a different dialysis center during the study, rendering follow-up per protocol, impractical.
* Patient is participating in, or has participated in, another study with an investigational drug within 30 days prior to signing the informed consent form.
* Women who are pregnant or lactating
* HIV positive (medical history review and patient report)
* Patient is on potent CYP3A4 Inhibitor or Inducer Drugs within one week of starting study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bolton, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited our subjects from 3 clinics at the University of Virginia. Our clinics were located at the Dialysis Units in Charlottesville, VA, Fisherville, VA, and Zion Crossroads, VA. Subjects were recruited into this study between March 2007 and August 2008.
Pre-assignment Details: 49 Subjects were recruited; 26 Subjects started intervention (4 Subjects started study intervention and then were dropped from the study), 22 Subjects Completed this trial. 1 Subject withdrew their consent prior to study intervention. 22 Subjects did not meet inclusion/exclusion criteria.
Groups:
- MK-0677 First, Then Placebo: Subjects took 25mg of MK-0677 for at least 30 Days.
- Placebo First, Then MK-0677: Subjects took Placebo for at least 30 days.
Period: First Intervention
Arm/Group | MK-0677 First, Then Placebo | Placebo First, Then MK-0677
Started | 17 | 9
Completed | 15 | 9
Not Completed | 2 | 0
Period: Washout Period for 30 Days
Arm/Group | MK-0677 First, Then Placebo | Placebo First, Then MK-0677
Started | 15 | 9
Completed | 13 | 9
Not Completed | 2 | 0
Period: Second Intervention
Arm/Group | MK-0677 First, Then Placebo | Placebo First, Then MK-0677
Started | 13 | 9
Completed | 13 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to placebo first and MK-0677 first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (14.4)
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in IGF-1 After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the IGF-1 levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: 22 Subjects completed both interventions and lab results were available.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- MK-0677: Subjects took 25mg of MK-0677 for at least 30 Days.
- Placebo: Subjects took Placebo for at least 30 days.
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 22
ng/ml | 92.7 (62.3) | 6.7 (40.2)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in IGF-1 is the same for both the MK-0677 and placebo interventions. Power calculation: We assumed that the IGF-I data will be lognormally distributed and thus the parameter of interest will be the IGF-1 geometric mean. If n=22 individuals complete the study and the intervention effect is 48% greater for one intervention than the other we will have at least 0.80 power to reject the null hypothesis; Test type: Superiority or Other; p < 0.001, ANCOVA — The IGF-1 data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

2. Secondary Outcome: Change in Acyl-Ghrelin After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the Acyl-Ghrelin levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention.
Population: 22 subjects completed both interventions.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 22
pg/ml | -23.4 (68.9) | 3.5 (150.3)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in Acyl-Ghrelin is the same for both the MK-0677 and placebo interventions. Because Acyl-Ghrelin is considered as a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.169, ANCOVA; The Acyl-Ghrelin data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

3. Secondary Outcome: Change in Leptin After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the Leptin levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: 22 subjects completed both interventions.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 22
ng/ml | 24.4 (50.2) | -6.9 (30.4)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in leptin is the same for both the MK-0677 and placebo interventions. Because Leptin is considered a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.063, ANCOVA; The Leptin data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

4. Secondary Outcome: Change in Insulin After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the Insulin levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: 22 subjects completed both interventions.
Measure: Mean (Standard Deviation); unit: uIU/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 22
uIU/ml | 3.77 (10.5) | -.2 (12.5)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in serum-insulin is the same for both the MK-0677 and placebo interventions. Because serum-insulin is considered a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.075, ANCOVA; The insulin data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

5. Secondary Outcome: Change in Des-Acyl Ghrelin After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the Des-Acyl Ghrelin levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: 22 Subjects completed both interventions.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 22
pg/ml | 30.2 (201.5) | -44.05 (157.4)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Test type: Superiority or Other; p = .782, ANCOVA

6. Secondary Outcome: Change in TNF-alpha After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the TNF-alpha levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: 22 subjects had samples available for the MK-0677 intervention, and 21 samples were available for the placebo intervention.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 21
pg/ml | 1.2 (5.9) | -0.7 (14.6)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in TNF-a is the same for both the MK-0677 and placebo interventions. Because Acyl-Ghrelin is considered as a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.385, ANCOVA; The TNF-a data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

7. Secondary Outcome: Change in CRPs After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the CRPs levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: 22 Subjects completed both interventions.
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 22
mg/ml | 2.6 (13.4) | 6.0 (32.7)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in CRPs is the same for both the MK-0677 and placebo interventions. Because CRPs is considered as a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.929, ANCOVA; The CRPs data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

8. Secondary Outcome: Change in IL-1 After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the IL-1 levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 21
pg/ml | 0.0 (0.2) | -0.0 (0.3)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in IL-1 is the same for both the MK-0677 and placebo interventions. Because IL-1 is considered as a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.905, ANCOVA; The IL-1 data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

9. Secondary Outcome: Changes in the Following Level: IL-6
Description: Change in IL-6 after 30 days of intervention.
Time Frame: After the subject has comleted their last visit
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 21
pg/mL | 3.1 (5.2) | 0.8 (6.9)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Test type: Superiority or Other; p = 0.233, ANCOVA

10. Secondary Outcome: Change in IL-10 After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the IL-10 levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 21
pg/ml | -0.1 (1.9) | 0.7 (1.7)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in IL-10 is the same for both the MK-0677 and placebo interventions. Because IL-10 is considered as a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.277, ANCOVA; The IL-10 data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

11. Secondary Outcome: Change in Esterase After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the Esterase levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: 22 subjects completed both interventions and results were available.
Measure: Mean (Standard Deviation); unit: units/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 22
units/ml | -1.6 (10.3) | -1.3 (12.6)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in esterase is the same for both the MK-0677 and placebo interventions. Because Acyl-Ghrelin is considered as a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.875, ANCOVA; The esterase data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

12. Secondary Outcome: Change in Adiponectin After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the Adiponectin levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 21
ng/ml | 1242.0 (7858.1) | 735.1 (4485.0)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in adiponectin is the same for both the MK-0677 and placebo interventions. Because Acyl-Ghrelin is considered as a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.545, ANCOVA; The adiponectin data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

13. Secondary Outcome: Change in Ghrelin After 30 Days of Intervention Compared to Baseline Level.
Description: Looking for a change in the Ghrelin levels after the subject has been on intervention for 30 days compared to baseline levels.
Time Frame: Baseline and after 30 days of intervention
Population: 22 subjects completed both interventions and lab results were available for all 22.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | MK-0677 | Placebo
Number analyzed (Participants) | 22 | 22
pg/ml | 6.9 (162.5) | -40.5 (192.5)
Statistical Analysis 1: Comparison: MK-0677 vs Placebo; Null hypothesis: the intra-subject pre-intervention to post-intervention change in Total-Ghrelin is the same for both the MK-0677 and placebo interventions. Because Acyl-Ghrelin is considered as a secondary outcome, no power analysis was conducted; Test type: Superiority or Other; p = 0.900, ANCOVA; Total ghrelin data were analyzed on the natural logarithmic scale via a linear mixed model in correspondence to a 2-period crossover design ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse Events were collect from the time the subject started the first intervention and ended two weeks from the last study visit.
Arm/Group | MK-0677 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/26 | 3/26
Other Adverse Events (participants affected / at risk) | 5/26 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0677 (N=26) | Placebo (N=26)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Clotted Permacath caused the renal failure
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Ischemic Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eroded Arteriovenous Dialysis Graft (Surgical and medical procedures) | 1 (1) | 0 (0) — Arteriovenous dialysis graft had eroded through the forearm skin which caused episodic pulsatile bleeding through the eroded graft.
Perm-A-Cath Line Infection (Infections and infestations) | 1 (1) | 0 (0) — Perm-A-Cath Line Infection that caused staphylococcus Epidermidis Bacteremia and Septic Deep Vein Thrombosis
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Hyperkalemia (Cardiac disorders) | 0 (0) | 1 (1)
Supratherapeutic INR (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0677 (N=26) | Placebo (N=26)
Cold, Cough, Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Nausea, Upset Stomach (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
We completed the appropriate number of subjects to get the statistical data needed. We had several screen fails (subjects that did not meet the inclusion/exclusion criteria.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No